CLINICAL TRIAL: NCT07398014
Title: The New Possibility of Treating Overactive Bladder With Radiofrequency - a Prospective, Randomized, Placebo Controlled (Single-blind) Clinical Trial
Brief Title: The New Possibility of Treating Overactive Bladder With Radiofrequency
Acronym: RF and OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Maribor (Other)
Responsible Party: Principal Investigator, Damir Franic, assist. prof. MD PhD, director, University Maribor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ginek dr franic
Record Dates: First submitted 2025-09-05; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Overactive Bladder and Urge Urinary Incontinence
Keywords: overactive bladder; urge urinary incontinence; radiofrequency treatment; quality of life
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: prospective randomized placebo control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency as the novel option for treating OAB and UUI (Placebo Comparator): We include 80 women with syptoms of OAb adn UUI, using validated q ICIQ-OAB, ICIQ-flutsex; ICIQ-OABQoL. Half of them were recruited in study group and half of them in placebo group. Follow-up was at 3,6 adn 12 months. That was the frist part of the study. After that we aplied RF for the women who were in placebo group with the same protocol
  Interventions: Device: radiofrequency - TECAR
- we aplied RF for the women who were in placebo group with the same protocol -"cross-over study" (Active Comparator)
  Interventions: Device: radiofrequency - TECAR

INTERVENTIONS:
Device: radiofrequency - TECAR — applied RF for 20 minutes with active probe oaver the bladder and pasive probe on the lumbar region. We applied 4 treatment 2 times/weekly

SUMMARY:
A prospective, randomized, single-blind, placebo-controlled study was conducted from June 2023 to May 2025. The study enrolled 95 women (N=48 in the study group; N=47 in the placebo group) who presented with confirmed symptoms of OAB and UUI prior to enrollment. Symptom severity and quality of life were assessed using validat-ed questionnaires from the International Consultation on Incontinence Questionnaires (ICIQ), specifically ICIQ-OAB, ICIQ-OABqol, and ICIQ-FLUTSsex. A higher score on these questionnaires indicated a worse quality of life, while a lower score indicated im-provement. Symptomatology was monitored at 3, 6, and 12 months post-RF applica-tion, at which points women completed all three validated questionnaires again. Prior to study commencement, all subjects provided informed consent. Before the initial RF treatment, urine analysis and urine culture were performed on all patients to rule out urinary infections. The study protocol was approved by the National Ethical Committee of the Republic of Slovenia (No.0120-184/2023-2711-15). The study was also submitted to Clinical Trials.gov (NCT 06080217), although it was not completed as RF is not yet an approved device for treating OAB.

2.1. Inclusion Criteria Women with clear signs of OAB who were not currently using pharmacological treatment (antimuscarinics/beta-3 agonists) were included. Patients who had previously used OAB medications but had discontinued them (due to side effects or ineffective-ness) at least 3 months prior to enrollment were also eligible for this study.

2.2. Exclusion Criteria Exclusion criteria included an inserted heart pacemaker, unexplained vaginal bleeding, inflammation of the vagina and/or uterus or uterine appendages, bacterial or viral infections (including urinary tract infections), impaired immune system, sclero-dermia, previous radiation treatment, or burns in the treatment area. Women with stress urinary incontinence (SUI) or mixed urinary incontinence (MUI) were also ex-cluded from this study. Patients were positioned in the lithotomy position with extended lower extremities. Probes were placed on the lower abdomen, in the bladder area (active probe), and on the lumbar spine (passive probe). A capacitive probe, operating in the "free treat-ment"/"power control" program, delivered high-frequency electricity to the bladder for 20 minutes at a frequency of 1.0 MHz. The energy output was limited to achieve a maximum temperature of 41 °C. Initially, a maximum energy of 75% and a frequency of 0.8 MHz were applied. These parameters were adjusted downward based on patient comfort regarding the amount of heat experienced. Subsequently, the power was re-duced to 50%, and the frequency was increased to 1.0 MHz, which resulted in moderate energy absorption. This energy level was maintained throughout the procedure, with patients absorbing an average of 18-19 kJ of energy.

The placebo (sham) group was also connected to the RF device, with an active probe placed on the bladder area and a passive probe on the lumbar area. The device was activated for 20 minutes but did not emit electricity. Patients in the placebo group were blinded to the fact that their energy had not been delivered. Following the study's conclusion, participants in the placebo group were informed of their random as-signment and were offered the active RF procedure.The primary endpoint was to confirm the statistically significant reduction in OAB and/or UUI symptoms observed in a prior pilot study. The secondary endpoint aimed to determine the optimal frequency for RF reapplication to achieve good Quality of Life (QoL) and maintain minimal symptomatologyPower analysis Based on literature data and our pilot study, we assume that the success rate for RF will be 60% and for placebo 25%. Considering these figures, we assume that we will need 30 patients for each group, but we must take into account the dropout during the study group, as well as in placebo gorup, so we included more patients per group in the study, so a total of 95 patients were included for randomization.

2.4.1. Statistics methods To assess the general characteristics of both groups, either the Student's t-test or the Mann-Whitney U test was employed, depending on data distribution.Statistical analy-sis was performed using generalized estimating equations (GEE) to account for the cor-relation of repeated measurements within subjects. A linear GEE model incorporating an identity link function and a Gaussian distribution was fitted. The primary predictors included time, group (study vs. control), and their interaction (time × group), with ad-ditional adjustment for the baseline covariate BMI. The interaction term was specifically included to evaluate whether the effect of time varied between the groups. Separate es-timates of the time effect within each group were derived by combining main and in-teraction effects, and their statistical significance was determined using z-tests.

DETAILED DESCRIPTION:
Frequency refers to the wavelength of the oscillation. Various frequencies are em-ployed in diathermy. Given that tissue absorption generally increases with frequency, it is often posited that lower frequencies yield better transfer efficiency. A frequency of 1 MHz has been proposed to effectively overcome cell membrane resistance and induce intracellular effects

. Power, or energy, is a fundamental component of electromag-netic fields. Electromagnetic waves transmit energy to a system through their electric and magnetic fields; greater field strength correlates with increased work capacity and higher energy transfer.

This energy desensitizes the bladder, thereby increasing its capacity, enhancing blood flow, and reducing the formation of free radicals, all of which contribute to im-proving the symptoms of OAB and UUI. Furthermore, the observation of an associated increase in the production of both epithelial and vascular growth factors-which pro-mote healing and angiogenesis, thereby augmenting blood circulation-offers a new perspective on this treatment.

Additionally, another mechanism by which high-power radiofrequency treats OAB and UUI involves a diathermic process. This process, generated by electromagnetic radiation, leads to an immediate retraction of existing collagen and subsequent activation of fibroblasts, ultimately resulting in non ablative neocollagenesis. Radiofrequency waves effectively penetrate to a depth sufficient to induce collagen production throughout the urethra, suggesting that these mechanisms can ameliorate OAB and UUI symptoms .

The RF application protocol employed in this study involved two weekly sessions of 20 minutes each, administered over a two-week period. Treatment efficacy was eval-uated by re-administering the questionnaires at 3, 6, and 12 . Randomization Method Randomization was conducted according to the guidelines of Fleiss , employ-ing a computer-generated sequence to allocate participants in a 1:1 ratio to either the in-tervention or control group. An independent statistician generated the allocation se-quence and had no involvement in participant enrollment.

post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* ICIQ-OAB criteria to determinate OAB

Exclusion Criteria:

* women with pacemaker, active malignancy, urinary infection, sclerodermia, active radioth., women with stress urinary incontinence, women who used pharmocological treatment for OAB less than 3 months before the RF, immunodeficiency

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
the influence of RF on OAB and UUI | the follow up was 3, 6 and 12 months, so the study was terminated after that period of time. For the QoL ICIQ-OABQol was used.A higher score on these questionnaires indicated a worse quality of life, while a lower score indicated improvement.
  to prove the efficacy of using RF in treating OAB and UUI in prospective randomized placebo control trial
number of participants with treatment is 95 divided in two groups- study and placebo related adverse events as assessed by CTCAEv4.o - there were NO adverse events the study satisfied the criteria of "Safety" change from baseline was reported in study g | from enrollment to the end of treatment at two weeks, then we repeat the symptomatology changes using validated questionnaires at 3-6-12 months
  A prospective, randomized, single-blind, placebo-controlled study was conducted from June 2023 to May 2025. The study enrolled 95 women (N=48 in the study group; N=47 in the placebo group) who presented with confirmed symptoms of OAB and UUI prior to enrollment. Symptom severity and quality of life were assessed using validated questionnaires from the International Consultation on Incontinence Questionnaires (ICIQ), specifically ICIQ-OAB, ICIQ-OABqol, and ICIQ-FLUTSsex. A higher score on these questionnaires indicated a worse quality of life, while a lower score indicated improvement. Symptomatology was monitored at 3, 6, and 12 months post-RF application, at which points women completed all three validated questionnaires again. Prior to study commencement, all subjects provided informed consent. Before the initial RF treatment, urine analysis and urine culture were performed on all patients to rule out urinary infections.
The primary endpoint was to confirm the statistically significant reduction in OAB and/or UUI symptoms observed in a prior pilot study | 3-6-12 months
  A higher score on these questionnaires indicated a worse symptomatology, while a lower score indicated improvement.
radiofrequency in treating overactive bladder and urge urinary incontinence | 3-6-12 months
  The primary endpoint was to confirm the statistically significant reduction in OAB and/or UUI symptoms observed in a prior pilot study.

SECONDARY OUTCOMES:
how many times needs to fullfill optimal QoL and cessation of symptoms | 3-6-12 months
  The secondary endpoint aimed to determine the optimal frequency for RF reapplication to achieve good Quality of Life (QoL) and maintain minimal symptomatology. A higher score on these questionnaires indicated a worse quality of life, while a lower score indicated improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Damir Franić, Rogaška Slatina, Slovenia

IPD SHARING:
Plan to Share IPD: No